CLINICAL TRIAL: NCT03213496
Title: Impact of a Routine of Pre-surgical Walk for Non Cardiac Adult Patients Compared to Conventional Intervention (Not Recommended Exercise) in Reducing the Length of Hospital Stay and the Time of Onset of Ambulation.
Brief Title: Promotion of Ambulation Before Non-cardiac Surgery
Acronym: PAMP-Phase2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Cardioinfantil Instituto de Cardiología (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CEIC-2224-2015
Record Dates: First submitted 2017-07-05; First posted 2017-07-11 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2017-07

CONDITIONS: Non-cardiac Surgery
Keywords: clinical trial, non cardiac surgery, walking.
MeSH Terms: interventions — Preoperative Exercise

STUDY DESIGN:
Intervention Model Description: Adult patients programmed for elective non-cardiac surgery, prior informed consent, will be randomized to an intervention (prescription of a programed walking) in the period of 2-3 weeks before surgery or will be assigned to a control group/conventional care.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Data of outcomes will be evaluated by statisticians.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Walk prescription (Experimental): Walk prescription for all weeks before non-cardiac surgery. Duration of walk must be of 30-40 minutes every day for five days at the week or until complete 150 minutes at the week, for all weeks up to the surgery.
  Interventions: Behavioral: Walk prescription
- Conventional care (Other): Currently patients do not receive exercise (walk)-prescription before non cardiac surgery.
  Interventions: Other: Conventional care

INTERVENTIONS:
Behavioral: Walk prescription — 30-40 minutes daily, for five days at the week, all weeks up to surgery.
  Other Names: prehabilitation
  Arms: Walk prescription
Other: Conventional care — Patient do not walk before surgery
  Arms: Conventional care

SUMMARY:
Primary Determine the impact of prescribing a routine pre-surgical walk scheduled compared to conventional intervention (not recommended exercise) in reducing the length of hospital stay and the time of onset of ambulation during postoperative hospitalization, in patients with ability to move, ≥30 years who will undergo non-cardiac surgery.

Secondary

1. Evaluate ischemic cardiovascular events (AMI), stroke (CVA) and cardiac mortality during hospitalization.
2. Evaluate the incidence of falls during hospitalization.

Methodology The PAMP project phase II, as a component of CARDIECOL program will be implemented by designing a pilot study, a randomized controlled trial. Adult-patients with greater than or equal to 30 years old entering elective non-cardiac surgery, prior informed consent will be randomized to an intervention prescribed of walking in the period of 2-3 weeks before surgery or will be assigned to a Control group/conventional care. The study was not blinded to patients, but evaluation and analysis of the data will be blinded for researchers and statisticians. Patients will be evaluated on their previous level of physical activity and will be evaluated by a physiatrist doctor for prescribing the walk (exercise). This study will include a sample of 500 patients, with capacity to mobilize, ability to walk at least 30 min/by day (150 min by week) for at least 1 week before surgery. Patients have to be hospitalized for at least 24 hours after the surgical procedure. Outcomes are length of stay, and time to first walk. Other results are evaluation falls during hospitalization and the presence of falls, report of cardiovascular events, and death by group.

Expected results

DETAILED DESCRIPTION:
Randomization was planned to be performed one to five weeks before non-cardiac surgery for all eligible patients, once they have decided to participate in the study. It was performed on a random computed to an intervention group (Walk prescription); or conventional care group (no exercise) in a 2:1 relation respectively. Intervention and Management Processes The pre surgical intervention walk routine is defined of at least 150-300 minutes of walk before going into surgery.

Analysis will be following the principle of intention to treat. A description of categorical and quantitative demographic data will be performed. Evaluation will also include the mean difference in the length of hospital stay for each of the groups and standard deviation, given a confidence interval of 95%. An analysis of the time of occurrence of the first walk using the Kaplan-Meier estimator will be performed.

ELIGIBILITY:
Inclusion Criteria:

* undergoing non-cardiac surgery
* general anesthesia or epidural or spinal anesthesia
* age ≥ 30 years
* able to walk and communicate

Exclusion Criteria:

* having any alteration of their state of consciousness
* altered mental status and communication

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Length of stay | Up 40 weeks in hospitalization
  Total stay hours

SECONDARY OUTCOMES:
Falls | Up 40 weeks in hospitalization
  Fall event reported in patients´ charts
Ischemic events | Up 40 weeks in hospitalization
  Myocardial infarction or stroke
Time to the first walk | Up 40 weeks in hospitalization
  First time out of the bed registered in patients´charts

CONTACTS AND LOCATIONS:
Overall Officials: Olga Cortés, PI, Principal Investigator — Fundación Cardioinfantil Instituto de Cardiología
Locations (2):
- Colombia (2):
  - Fundación CardioInfantil Instituto de Cardiología, Bogotá, Cundinamarca
  - Clinica Carlos Ardila Lulle-FOSCAL, Bucaramanga, Santander Department

IPD SHARING:
Plan to Share IPD: No
Data will be registered in indepenedent filles in folders; and also data will be typed on the PAMP Data base (CARDIECOL). Data can be monitored by a coordinator.

REFERENCES:
- [Background] Carli F, Charlebois P, Stein B, Feldman L, Zavorsky G, Kim DJ, Scott S, Mayo NE. Randomized clinical trial of prehabilitation in colorectal surgery. Br J Surg. 2010 Aug;97(8):1187-97. doi: 10.1002/bjs.7102. PMID 20602503
- [Background] Santa Mina D, Scheede-Bergdahl C, Gillis C, Carli F. Optimization of surgical outcomes with prehabilitation. Appl Physiol Nutr Metab. 2015 Sep;40(9):966-9. doi: 10.1139/apnm-2015-0084. Epub 2015 May 13. PMID 26300015
- [Background] Mayo NE, Feldman L, Scott S, Zavorsky G, Kim DJ, Charlebois P, Stein B, Carli F. Impact of preoperative change in physical function on postoperative recovery: argument supporting prehabilitation for colorectal surgery. Surgery. 2011 Sep;150(3):505-14. doi: 10.1016/j.surg.2011.07.045. PMID 21878237
- [Derived] Cortes OL, Herrera-Galindo M, Becerra C, Rincon-Roncancio M, Povea-Combariza C, Esparza-Bohorquez M. Preoperative walking recommendation for non-cardiac surgery patients to reduce the length of hospital stay: a randomized control trial. BMC Sports Sci Med Rehabil. 2021 Jul 28;13(1):80. doi: 10.1186/s13102-021-00317-w. PMID 34321092